CLINICAL TRIAL: NCT05652322
Title: A Randomized Trial Comparing Prolonged Intravenous Therapy Versus Early Initiation of an Oral Loop Diuretic in Patients Hospitalized for Decompensated Chronic Heart Failure
Brief Title: Prolonged Intravenous Therapy Versus Early Initiation of an Oral Loop Diuretic in Decompensated Heart Failure
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: no recruitment
Sponsor: Jan Kochanowski University (Other)
Responsible Party: Principal Investigator, Zbigniew Siudak, Professor, Jan Kochanowski University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1/KCW/2022
Record Dates: First submitted 2022-12-07; First posted 2022-12-15 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Heart Failure
Keywords: diuretic; oral; intravenous
MeSH Terms: conditions — Heart Failure | interventions — Furosemide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group 1 (Active Comparator): prolonged intravenous loop diuretic treatment - furosemide
  Interventions: Drug: Furosemide Injection
- Group 2 (Experimental): Early (48 hrs) change to oral loop diuretic - furosemide - 150% eqivalent iv dose
  Interventions: Drug: Furosemide Pill 150% equivalent iv dose
- Group 3 (Experimental): Early (48 hrs) change to oral loop diuretic - furosemide - 200% eqivalent iv dose
  Interventions: Drug: Furosemide Pill 200% equivalent iv dose

INTERVENTIONS:
Drug: Furosemide Pill 150% equivalent iv dose — change from intravenous to oral furosemide
  Arms: Group 2
Drug: Furosemide Pill 200% equivalent iv dose — change from intravenous to oral furosemide
  Arms: Group 3
Drug: Furosemide Injection — change from intravenous to oral furosemide
  Arms: Group 1

SUMMARY:
The goal of this clinical study is to compare treatment regimens of loop diuretics in patients with decompensated heart failure. The main aim is to answer if early change from intravenous to oral loop diuretics is safe and effective.

ELIGIBILITY:
Inclusion Criteria:

* Patient hospitalized due to exacerbation of heart failure symptoms, where AHF is the main cause of hospitalization. To be included in the study, all criteria 1 to 6 must be met:

  1. Fluid Retention Features:

     * Described congestion above the lung fields on chest X-ray
     * rales on chest auscultation
     * Peripheral edema, yielding to pressure occurring within the limbs or the sacral part of the spine
     * Increased pressure in the jugular veins (>=8 cm H2O)
  2. The concentration of natiuretic peptides must be assessed within 24 hours of admission to the hospital and be:

     ✔ NTpro-BNP >450 pg/mL for <55 years, 900 pg/mL for 55-75 years, and >1800 pg/mL for >75 years
  3. Exacerbation of heart failure treated with at least 40 mg of furosemide IV. (or 20 mg torasemide equivalent)
  4. Left ventricular ejection fraction < 50% (assessed and documented in the last 12 months prior to study entry)
  5. Age >= 18 years
  6. The study participant gave and signed an informed consent to participate in the study. No medical procedure related to the study was performed prior to giving informed consent.

Exclusion Criteria:

* 1. Shortness of breath caused by respiratory infection, exacerbation of bronchial asthma, COPD 2. Body temperature > 38 C, signs of active infection requiring antibiotic therapy, sepsis, infective endocarditis 3. An episode of acute coronary syndrome, stroke or TIA within 6 months before randomization 4. Severe valvular disease requiring or in the process of qualifying for repair 5. Patients requiring dialysis (in the past, during hospitalization or in the process of qualifying for dialysis) 6. History of alcohol abuse in the last 2 years before randomization 7. Pregnancy or breastfeeding 8. Active cancer or in remission for less than 5 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-12-07 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
number of patients requiring hospitalization | 12 weeks
  any hospitalization due to cardiovascular reasons
Time to hospitalization measured in days | Up to 12 weeks
  Time to any hospitalization due to cardiovascular reasons

SECONDARY OUTCOMES:
Death | 12 weeks
  Cardiovascular death
New York Heart Association NYHA class | 6 and12 weeks
  NYHA class assessment
assessment of quality of life | 12 weeks
  QoL by Minnesota questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Janusz Sielski, MD, PhD, Principal Investigator — Jan Kochanowski Univeristy in Kielce
Locations (3):
- Poland (3):
  - Wojewodzki Szpital Zespolony Klinika Nefrologii, Kielce
  - Wojewódzki Szpital Zespolony OIOK, Kielce
  - Wojewódzkie Wielospecjalistyczne Centrum Onkologii i Traumatologii im. M. Kopernika, Oddzial Kardiologii, Lodz

REFERENCES:
- See also: Jan Kochanowski University Kielce, Poland — https://interna.ujk.edu.pl/